CLINICAL TRIAL: NCT01544166
Title: Open-label, Multicenter, Pharmacokinetic, and Safety Study in Children (Term Newborn Infants to 23 Months of Age) Undergoing a Contrast-enhanced MRI With an Intravenous Injection of 0.1 mmol/kg BW Gadobutrol 1.0 M
Brief Title: Gadobutrol Pharmacokinetic and Safety Study in Pediatric Subjects Aged <2 Years (Term Newborn Infants to Toddlers 23 Months of Age Inclusive)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91741; 2010-023003-96 (EudraCT Number)
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Magnetic Resonance Imaging
Keywords: Gadolinium, Pediatrics, MRI, contrast
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall study (Experimental)
  Interventions: Drug: Gadobutrol (Gadavist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, BAY86-4875) — Single intravenous bolus injection of gadobutrol 0.1 mmol/kg BW in term newborns to infants <2 years of age.

SUMMARY:
The main purpose of this study is to collect data on the way gadobutrol is taken into, moves around, and is eliminated from, the body of children aged 0 to less than 2 years. The study will also evaluate safety and tolerability, and efficacy of gadobutrol.

A maximum total amount of approximately 5 ml of blood will be needed for these analyses which will be drawn within 2-3 days.

Gadobutrol is a contrast agent used for enhancement of Magnetic Resonance Imaging (MRI), potentially allowing better visibility of tissues in the body. Children aged under 2 years scheduled for a routine contrast-enhanced MRI examination of any body region may take part in this study, in which case they will receive gadobutrol as contrast agent intravenously at the standard dose of 0.1 mmol/kg (0.1 ml/Kg) of body weight. Only subjects without renal insufficiency of any intensity (i.e. estimated Glomerular Filtration Rate <80% of age adjusted normal value calculated based on the Schwartz formula) will be included in the trial.

The duration of this study as a whole is around 1 year and the total number of children to be enrolled is 50. A child will be expected to take part in the study for around 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects aged <2 years (term newborn infants to toddlers 23 months of age inclusive)
* Subject is scheduled to undergo routine gadolinium-enhanced MRI of any body region

Exclusion Criteria:

* Subjects undergoing a change in chemotherapy within 48 hours prior to and up to 24 hours after gadobutrol injection
* Any planned intervention during the study and up to 24 hours after gadobutrol injection (excluding lumbar puncture)
* Subjects who received or will receive any investigational product within 48 hours before gadobutrol injection or during study participation
* Subjects who received or will receive any other contrast agent within 48 hours prior to gadobutrol injection or up to 24 hours after gadobutrol injection
* Subjects with contraindication for MRI such as iron metal implants (e.g. aneurysm clips)
* History of anaphylactoid or anaphylactic reaction to any allergen including drugs and contrast agents
* Subject with renal insufficiency of any intensity, i.e. estimated Glomerular Filtration Rate <80% of age adjusted normal value calculated based on the Schwartz formula

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2013-11-28 (Actual); Study Completion 2013-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (5):
  - Savannah, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Houston, Texas
- Edmonton, Alberta, Canada
- Germany (3):
  - Dresden, Saxony
  - Halle, Saxony-Anhalt
  - Jena, Thuringia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=91741&attachmentIdentifier=6a1fb590-4050-4a4c-84fb-8bea151dcd1f&fileName=91741_study_synopsis_CTP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric subjects who were less than (<) 2 years of age, scheduled to undergo contrast-enhanced magnetic resonance imaging (MRI) for routine diagnostic purposes were included in the study and were recruited from 9 centres in Canada, Germany and United States of America.
Pre-assignment Details: Total of 47 subjects were screened worldwide in the study and 44 were enrolled (i.e. assigned to study drug). It included 3 screening failures (3 patients were not treated and did not complete the study).
Groups:
- Overall Study: Single intravenous bolus injection of gadobutrol 0.1 mmol/kg BW in term newborns to infants <2 years of age.
Period: Overall Study
Arm/Group | Overall Study
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: months] | 8.8 (7.1)
Age, Customized [Number; unit: Participants]
  Newborns (0-27 days) | 5
  Infants and toddlers (28 days-23 months) | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to Infinity of Gadobutrol: Individual
Description: AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC from time 0 (start of injection) to infinity was reported in micromole*hour per liter (micromole*h/L).
Time Frame: Blood samples were collected at 3 timepoints between 15 minutes and 8 hours post administration of gadobutrol
Population: Per-protocol set (PPS) included those subjects who received the appropriate dose of gadobutrol based on the dose specification of 0.1 mmol/kg BW plus/minus 10% and had quantifiable gadolinium plasma concentrations in at least 1 valid PK sample.
Measure: Median (Full Range); unit: micromole*h/L
Arm/Group | Overall Study
Number analyzed (Participants) | 43
micromole*h/L | 776 [544 to 1470]

2. Primary Outcome: Body Weight-Normalized Total Body Clearance (CL) of Gadobutrol From Plasma: Individual
Description: Clearance is the volume of the fluid presented to the eliminating organ that is effectively completely cleared of drug per unit time and depends on the rate of elimination. CL of gadobutrol normalized for body weight, was reported in Liter per hour per kilogram (L/(h*kg).
Time Frame: Blood samples were collected at 3 timepoints between 15 minutes and 8 hours post administration of gadobutrol
Population: PPS included those subjects who received the appropriate dose of gadobutrol based on the dose specification of 0.1 mmol/kg BW plus/minus 10% and had quantifiable gadolinium plasma concentrations in at least 1 valid PK sample.
Measure: Median (Full Range); unit: L/(h*kg)
Arm/Group | Overall Study
Number analyzed (Participants) | 43
L/(h*kg) | 0.128 [0.0666 to 0.184]

3. Primary Outcome: Body Weight-Normalized Apparent Volume of Distribution at Steady State (Vss) of Gadobutrol in Plasma: Individual
Description: Vss is an estimate of drug distribution independent of the elimination process and is proportional to the amount of drug in the body versus the drug plasma concentration at steady-state.
Time Frame: Blood samples were collected at 3 timepoints between 15 minutes and 8 hours post administration of gadobutrol
Population: as for outcome 2
Measure: Median (Full Range); unit: L/kg
Arm/Group | Overall Study
Number analyzed (Participants) | 43
L/kg | 0.277 [0.236 to 0.409]

4. Primary Outcome: Mean Residence Time (MRT) of Gadobutrol in Plasma: Individual
Description: MRT is the average time that the molecules introduced into the body stay in the body. MRT of Gadobutrol is expressed in hours.
Time Frame: Blood samples were collected at 3 timepoints between 15 minutes and 8 hours post administration of gadobutrol
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Overall Study
Number analyzed (Participants) | 43
hours | 2.18 [1.57 to 4.68]

5. Primary Outcome: Terminal Elimination Half-Life (t1/2) of Gadobutrol From Plasma: Individual
Description: Half-life refers to the elimination of the drug, that is, the time it takes for the blood plasma concentration to reach half the concentration. Terminal elimination half-life of gadobutrol from plasma is expressed in hours and is derived from the terminal slope of the concentration versus time curve.
Time Frame: Blood samples were collected at 3 timepoints between 15 minutes and 8 hours post administration of gadobutrol
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Overall Study
Number analyzed (Participants) | 43
hours | 1.62 [1.16 to 3.37]

6. Primary Outcome: Simulation of Plasma Concentration of Gadobutrol at 20 Minutes Post-Injection (C20)
Description: Simulation is the use of the model to predict data other than observed data, in this case early Gadobutrol plasma concentration after intravenous injection. Plasma concentration serves as a surrogate for efficacy (signal and contrast enhancement) in MRI. C20 was simulated for virtual pediatric subjects with homogenous distribution over age. Simulated median (5th and 95th percentile in parenthesis) gadolinium plasma concentrations for a dose of 0.1 mmol/kg body weight were presented.
Time Frame: 20 minutes post-injection
Population: PPS included those subjects who received the appropriate dose of gadobutrol based on the dose specification of 0.1 mmol/kg BW plus/minus 10% and had quantifiable gadolinium plasma concentrations in at least 1 valid PK sample. Here number of subjects analysed= 43. C20 was simulated for 2400 virtual paediatric participants.
Measure: Median (Full Range); unit: micromole/L
Arm/Group | Overall Study
Number analyzed (Participants) | 43
micromole/L | 339 [230 to 456]

7. Primary Outcome: Simulation of Plasma Concentration of Gadobutrol at 30 Minutes Post-Injection (C30)
Description: Simulation is the use of the model to predict data other than observed data, in this case early Gadobutrol plasma concentration after intravenous injection. Plasma concentration serves as a surrogate for efficacy (signal and contrast enhancement) in MRI. C30 was simulated for virtual pediatric subjects with homogenous distribution over age. Simulated median (5th and 95th percentile in parenthesis) gadolinium plasma concentrations for a dose of 0.1 mmol/kg body weight were presented.
Time Frame: 30 minutes post-injection
Population: PPS included those subjects who received the appropriate dose of gadobutrol based on the dose specification of 0.1 mmol/kg BW plus/minus 10% and had quantifiable gadolinium plasma concentrations in at least 1 valid PK sample. C30 was simulated for 2400 virtual paediatric participants.
Measure: Median (Full Range); unit: micromole/L
Arm/Group | Overall Study
Number analyzed (Participants) | 43
micromole/L | 292 [194 to 394]

8. Secondary Outcome: Number of Subjects With Anatomical Area Evaluated
Description: Subjects were referred for MRI of any body region. The primary anatomical area to be evaluated by MRI was assessed. Anatomical Area was recorded prior to gadobutrol injection for the unenhanced MRI procedure and after gadobutrol injection for the gadobutrol-enhanced MRI procedure. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: Full analysis set (FAS) included all subjects who had combined unenhanced and enhanced image sets available regardless of any other protocol deviation.
Measure: Number; unit: subjects
Groups:
- Unenhanced MRI Assessment: Assessment was provided for the unenhanced image set alone in all FAS subjects.
- Combined MRI Assessment: Assessment was provided for the combined unenhanced and enhanced image set in all FAS subjects.
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: Liver | 1 | 1
  Brain: Brain | 20 | 20
  Brain: Orbit and brain | 1 | 1
  Chest/thorax: Lung | 2 | 2
  Head/neck: Head | 3 | 3
  Head/neck: Neck | 1 | 1
  Head/neck: Skull base/mandible | 1 | 1
  Lymphatic system: Right arm | 1 | 1
  Pelvic area:Trochanter major, femur neck | 1 | 1
  Pelvic area: Testis | 1 | 1
  Retroperitoneal: Kidney | 6 | 6
  Retroperitoneal: Adrenal gland | 1 | 1
  Spine: Spinal cord | 4 | 4
  Spine: Lumbar spine | 1 | 1

9. Secondary Outcome: Number of Subjects With Technical Adequacy for Diagnosis
Description: The technical adequacy of the unenhanced image set and the combined unenhanced and enhanced image set was assessed based on the following 4 point scale: 1=Region visualized with artifacts compromising quality and interpretability of images, 2=Only partial evaluation of images possible, region not covered adequately anatomically, 3=Region visualized with artifacts, partially compromising image quality but evaluation and diagnosis still possible, 4=Region clearly visualized, excellent quality. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Score = 1 | 0 | 0
  Score = 2 | 0 | 0
  Score = 3 | 4 | 3
  Score = 4 | 40 | 41

10. Secondary Outcome: Number of Subjects With Technical Adequacy for Diagnosis by Body Region
Description: The technical adequacy of the the unenhanced image set and the combined unenhanced and enhanced image set was assessed based 4-point scale and body region. Four-point scale: 1=Region visualized with artifacts compromising quality and interpretability of images, 2=Only partial evaluation of images possible, region not covered adequately anatomically, 3=Region visualized with artifacts, partially compromising image quality but evaluation and diagnosis still possible, 4=Region clearly visualized, excellent quality. Evaluation was done on pre-injection and combined images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: Score 4 | 1 | 1
  Brain: Score 3 | 1 | 1
  Brain: Score 4 | 20 | 20
  Chest/thorax: Score 4 | 2 | 2
  Head/neck: Score 3 | 1 | 1
  Head/neck: Score 4 | 4 | 4
  Lymphatic system: Score 4 | 1 | 1
  Pelvic area: Score 4 | 2 | 2
  Retroperitoneal area: Score 4 | 7 | 7
  Spine: Score 3 | 2 | 1
  Spine: Score 4 | 3 | 4

11. Secondary Outcome: Number of Subjects by Overall Contrast Quality
Description: A qualitative assessment of the overall contrast using the following pre-defined 5-point scale: 1= None (for example, in case of a non-enhancing vessel), 2= Poor, 3= Moderate, 4= Good, 5= Excellent, was done. This parameter was assessed in the postcontrast MRI only, which is evaluated together with the unenhanced, this is why it is called combined. Data for combined MRI set was reported.
Time Frame: Images were taken post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Combined MRI Assessment
Number analyzed (Participants) | 44
subjects
  None | 1
  Poor | 0
  Moderate | 0
  Good | 5
  Excellent | 38

12. Secondary Outcome: Number of Subjects by Overall Contrast Quality by Body Region
Description: A qualitative assessment of the overall contrast using the following pre-defined 5-point scale: 1= None (for example, in case of a non-enhancing vessel), 2= Poor, 3= Moderate, 4= Good, 5= Excellent, was done in the postcontrast MRI only, which is evaluated together with the unenhanced, this is why it is called combined. Data for combined MRI set was reported.
Time Frame: Images were taken post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Combined MRI Assessment
Number analyzed (Participants) | 44
subjects
  Abdomen: Excellent | 1
  Brain: Good | 2
  Brain: Excellent | 19
  Chest/Thorax: Good | 1
  Chest/Thorax: Excellent | 1
  Head/Neck: Excellent | 5
  Lymphatic system: Excellent | 1
  Pelvic area: Excellent | 2
  Retroperitoneal: None | 1
  Retroperitoneal: Good | 1
  Retroperitoneal: Excellent | 5
  Spine: Good | 1
  Spine: Excellent | 4

13. Secondary Outcome: Number of Subjects With Presence of Pathology
Description: Presence of pathology was assessed for unenhanced and combined MRI sets and recorded as "yes/no". The number of lesions identified for each MRI set was recorded.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Yes | 33 | 33
  No | 11 | 11

14. Secondary Outcome: Number of Subjects With Presence of Pathology by Body Region
Description: Presence of pathology was assessed for unenhanced and combined MRI sets and recorded as "yes/no". The number of lesions identified for each MRI set was recorded. Results per body region were reported.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: No | 0 | 0
  Abdomen: Yes | 1 | 1
  Brain: No | 10 | 10
  Brain: Yes | 11 | 11
  Chest/Thorax: No | 0 | 0
  Chest/Thorax: Yes | 2 | 2
  Head/Neck: No | 0 | 0
  Head/Neck: Yes | 5 | 5
  Lymphatic system: No | 0 | 0
  Lymphatic system: Yes | 1 | 1
  Pelvic area: No | 0 | 0
  Pelvic area: Yes | 2 | 2
  Retroperitoneal: No | 0 | 0
  Retroperitoneal: Yes | 7 | 7
  Spine: No | 1 | 1
  Spine: Yes | 4 | 4

15. Secondary Outcome: Number of Subjects With Number of Lesions Detected
Description: Presence of pathology included presence of lesions and was recorded as "yes/no". If "yes" the number of subjects with specified lists of lesions and body region was reported. Evaluation was done on pre- injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: Full analysis set (FAS) included all subjects who had combined unenhanced and enhanced image sets available regardless of any other protocol deviation. 44 subjects in the FAS were analyzed. The number of subjects with presence of pathology was 33.
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Number of lesions=missing | 2 | 1
  Number of lesions=1 | 29 | 29
  Number of lesions=2 | 2 | 2
  Number of lesions=10 | 0 | 1

16. Secondary Outcome: Number of Subjects With Number of Lesions Detected by Body Region
Description: Presence of pathology included presence of lesions and was recorded as "yes/no". If "yes" the number of subjects with specified lists of lesions and body region was reported. Evaluation was done on pre- injection and combined (pre- and post-injection) images. Data of subjects with missing number of lesions or at least one lesion in unenhanced and combined MRI sets were reported.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 15
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: Missing lesion | 1 | 1
  Brain: 1 lesion | 10 | 10
  Brain: 2 lesion | 1 | 1
  Chest/Thorax: 1 lesion | 2 | 2
  Head/Neck: Missing lesion | 1 | 0
  Head/Neck: 1 lesion | 4 | 4
  Head/Neck: 10 lesion | 0 | 1
  Lymphatic system: 1 lesion | 1 | 1
  Pelvic area: 1 lesion | 2 | 2
  Retroperitoneal: 1 lesion | 6 | 6
  Retroperitoneal: 2 lesion | 1 | 1
  Spine: 1 lesion | 4 | 4

17. Secondary Outcome: Contrast Enhancement in Lesion or Vessel
Description: The contrast-enhancement for each lesion or vessel was recorded on a 4-point scale: 1 = None, lesion or vessel is not enhanced; 2 = Moderate, lesion or vessel is weakly enhanced; 3 = Good, lesion or vessel is clearly enhanced; 4 = Excellent, lesion or vessel is clearly and brightly enhanced. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  None | 44 | 3
  Moderate | 0 | 0
  Good | 0 | 6
  Excellent | 0 | 35

18. Secondary Outcome: Contrast Enhancement in Lesion or Vessel by Body Region
Description: The contrast-enhancement for each lesion or vessel was recorded on a 4-point scale: 1 = None, lesion or vessel is not enhanced; 2 = Moderate, lesion or vessel is weakly enhanced; 3 = Good, lesion or vessel is clearly enhanced; 4 = Excellent, lesion or vessel is clearly and brightly enhanced. Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: None | 1 | 1
  Blood vessel: None | 2 | 0
  Blood vessel: Excellent | 0 | 2
  Brain: None | 19 | 0
  Brain: Good | 0 | 1
  Brain: Excellent | 0 | 18
  Chest/Thorax: None | 2 | 1
  Chest/Thorax: Good | 0 | 1
  Head/Neck: None | 5 | 0
  Head/Neck: Good | 0 | 1
  Head/Neck: Excellent | 0 | 4
  Lymphatic system: None | 1 | 0
  Lymphatic system: Excellent | 0 | 1
  Pelvic area: None | 2 | 0
  Pelvic area: Good | 0 | 2
  Retroperitoneal: None | 7 | 1
  Retroperitoneal: Excellent | 0 | 6
  Spine: None | 5 | 0
  Spine: Good | 0 | 1
  Spine: Excellent | 0 | 4

19. Secondary Outcome: Number of Subjects With Border Delineation of Lesion of Vessel
Description: The border delineation for each lesion or vessel was recorded on a 4-point scale: 1 = None, no or unclear delineation of the boundary between the lesion or vessel and the surrounding tissue; 2 = Moderate, some aspects of border delineation covered; 3 = Good, almost clear delineation, but not complete on relevant slices; 4 = Excellent, clear and complete delineation.Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  None | 5 | 1
  Moderate | 6 | 0
  Good | 9 | 1
  Excellent | 24 | 42

20. Secondary Outcome: Number of Subjects With Border Delineation of Lesion of Vessel by Body Region
Description: The border delineation for each lesion or vessel was recorded on a 4-point scale: 1 = None, no or unclear delineation of the boundary between the lesion or vessel and the surrounding tissue; 2 = Moderate, some aspects of border delineation covered; 3 = Good, almost clear delineation, but not complete on relevant slices; 4 = Excellent, clear and complete delineation.The results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: Excellent | 1 | 1
  Blood vessel: Excellent | 2 | 2
  Brain: Moderate | 3 | 0
  Brain: Good | 6 | 0
  Brain: Excellent | 10 | 19
  Chest/Thorax: Good | 1 | 0
  Chest/Thorax: Excellent | 1 | 2
  Lymphatic system: Excellent | 1 | 1
  Pelvic area: Moderate | 1 | 0
  Pelvic area: Excellent | 1 | 2
  Retroperitoneal: None | 3 | 1
  Retroperitoneal: Excellent | 4 | 6
  Spine: None | 2 | 0
  Spine: Moderate | 2 | 0
  Spine: Excellent | 1 | 5
  Head/Neck: Good | 2 | 1
  Head/Neck: Excellent | 3 | 4

21. Secondary Outcome: Number of Subjects by Visualization of Lesion-Internal Morphology or Homogeneity of Vessel Enhancement
Description: The degree of visualization of internal morphology and structure was recorded on a 3-point scale: 1= Poor, the structure and internal morphology of the lesion or vessel is poorly visible; 2 = Moderate, the structure and internal morphology of the lesion or vessel is visible but sufficient information cannot be obtained; 3 = Good, the structure and internal morphology of the lesion or vessel is sufficiently visible for diagnostic purposes.Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Poor | 6 | 1
  Moderate | 11 | 0
  Good | 27 | 43

22. Secondary Outcome: Number of Subjects by Visualization of Lesion-Internal Morphology or Homogeneity of Vessel Enhancement by Body Region
Description: The degree of visualization of internal morphology and structure was recorded on a 3-point scale: 1 = Poor, the structure and internal morphology of the lesion or vessel is poorly visible; 2 = Moderate, the structure and internal morphology of the lesion or vessel is visible but sufficient information cannot be obtained; 3 = Good, the structure and internal morphology of the lesion or vessel is sufficiently visible for diagnostic purposes. Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: Good | 1 | 1
  Blood vessel: Good | 2 | 2
  Brain: Poor | 1 | 0
  Brain: Moderate | 5 | 0
  Brain: Good | 13 | 19
  Chest/Thorax: Moderate | 1 | 0
  Chest/Thorax: Good | 1 | 2
  Head/Neck: Poor | 1 | 0
  Head/Neck: Good | 4 | 5
  Lymphatic system: Good | 1 | 1
  Pelvic area: Moderate | 2 | 0
  Pelvic area: Good | 0 | 2
  Retroperitoneal: Poor | 3 | 1
  Retroperitoneal: Good | 4 | 6
  Spine: Poor | 1 | 0
  Spine: Moderate | 3 | 0
  Spine: Good | 1 | 5

23. Secondary Outcome: Number of Subjects With Diagnoses
Description: The following diagnoses were reported for both the unenhanced MRI and the combined MRI image sets: Other diagnoses, No lesions/normal, Congenital disease/syndrome, Malignant lesion, Inflammation, Structural malformation, Benign lesion, and Vascular malformation. Evaluation was done on pre- injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Benign lesion | 1 | 2
  Malignant lesion | 4 | 4
  Vascular malformation | 1 | 1
  Structural malformation | 2 | 2
  Inflammation | 2 | 3
  Congenital disease / syndrome | 6 | 8
  No lesion/Normal | 10 | 11
  Other | 18 | 13

24. Secondary Outcome: Number of Subjects With Diagnoses by Body Region
Description: The following diagnoses were reported for both the unenhanced MRI and the combined MRI image sets: Other diagnoses, No lesions/normal, Congenital disease/syndrome, Malignant lesion, Inflammation, Structural malformation, Benign lesion, and Vascular malformation. Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: Other | 1 | 1
  Brain: Malignant lesion | 1 | 1
  Brain: Inflammation | 1 | 1
  Brain: Congenital disease/syndrome | 3 | 3
  Brain: No lesion/Normal | 9 | 10
  Brain: Other | 7 | 6
  Chest/Thorax: Structural malformation | 1 | 1
  Chest/Thorax: Other | 1 | 1
  Head/Neck: Benign lesion | 1 | 1
  Head/Neck: Malignant lesion | 1 | 1
  Head/Neck: Inflammation | 1 | 1
  Head/Neck: Other | 2 | 2
  Lymphatic system: Vascular malformation | 1 | 1
  Pelvic area: Benign lesion | 0 | 1
  Pelvic area: Inflammation | 0 | 1
  Pelvic area: Other | 2 | 0
  Retroperitoneal: Malignant lesion | 1 | 1
  Retroperitoneal: Congenital disease/syndrome | 3 | 5
  Retroperitoneal: Other | 3 | 1
  Spine: Malignant lesion | 1 | 1
  Spine: Structural malformation | 1 | 1
  Spine: No lesion/Normal | 1 | 1
  Spine: Other | 2 | 2

25. Secondary Outcome: Number of Subjects With Additional Diagnostic Gain
Description: Additional diagnostic gain by the contrast-enhanced image set was assessed on a 3-point scale: scale 1 = Initial diagnosis unchanged, scale 2 = Initial diagnosis changed - improved, i.e. more specific, and scale 3 = Initial diagnosis changed -new diagnosis. Evaluation was done on combined (pre- and post- injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Combined MRI Assessment
Number analyzed (Participants) | 44
subjects
  Scale 1 | 19
  Scale 2 | 24
  Scale 3 | 1

26. Secondary Outcome: Number of Subjects With Additional Diagnostic Gain by Body Region
Description: Additional diagnostic gain by the contrast-enhanced image set was assessed on a 3-point scale: scale 1 = Initial diagnosis unchanged, scale 2 = Initial diagnosis changed - improved, i.e. more specific, and scale 3 = Initial diagnosis changed -new diagnosis. Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Combined MRI Assessment
Number analyzed (Participants) | 44
subjects
  Abdomen: Scale 2 | 1
  Brain: Scale 1 | 11
  Brain: Scale 2 | 9
  Brain: Scale 3 | 1
  Chest/Thorax: Scale 2 | 2
  Head/Neck: Scale 1 | 3
  Head/Neck: Scale 2 | 2
  Lymphatic system: Scale 2 | 1
  Pelvic area: Scale 2 | 2
  Retroperitoneal: Scale 1 | 3
  Retroperitoneal: Scale 2 | 4
  Spine: Scale 1 | 2
  Spine: Scale 2 | 3

27. Secondary Outcome: Number of Subjects With Confidence in Diagnosis
Description: Diagnostic confidence based on the unenhanced MRI image sets and thereafter on the combined MRI image sets were assessed on a 3-point scale, as 1 = Not confident, 2 = Confident and 3 = Very confident. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Not confident | 6 | 1
  Confident | 14 | 3
  Very confident | 24 | 40

28. Secondary Outcome: Number of Subjects With Confidence in Diagnosis by Body Region
Description: Diagnostic confidence based on the unenhanced MRI image sets and thereafter on the combined MRI image sets were assessed on a 3-point scale, as 3 = Very confident, 2 = Confident, and 1 = Not confident. Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Unenhanced MRI Assessment | Combined MRI Assessment
Number analyzed (Participants) | 44 | 44
subjects
  Abdomen: Confident | 1 | 1
  Brain: Not confident | 1 | 0
  Brain: Confident | 8 | 0
  Brain: Very confident | 12 | 21
  Chest/Thorax: Confident | 1 | 0
  Chest/Thorax: Very confident | 1 | 2
  Head/Neck: Confident | 2 | 0
  Head/Neck: Very confident | 3 | 5
  Lymphatic system: Very confident | 1 | 1
  Pelvic area: Not confident | 2 | 0
  Pelvic area: Confident | 0 | 2
  Retroperitoneal: Not confident | 3 | 1
  Retroperitoneal: Very confident | 4 | 6
  Spine: Confident | 2 | 0
  Spine: Very confident | 3 | 5

29. Secondary Outcome: Number of Subjects With Final Diagnosis
Description: The final diagnosis of the subjects was based on all clinical information available and was provided separately within 4 weeks after MRI. Evaluation was done on pre-injection and combined (pre- and post- injection) images.
Time Frame: Up to 4 weeks post-injection
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  Other diagnoses | 24
  Congenital disease/syndrome | 6
  No lesions/normal | 6
  Malignant lesions | 4
  Benign lesions | 2
  Infectious disease | 1
  Structural malformation | 1

30. Secondary Outcome: Number of Subjects With Final Diagnosis by Body Region
Description: The final diagnosis of the subjects was based on all clinical information available and was provided separately within 4 weeks after MRI. Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images. Only subjects with final diagnosis were reported.
Time Frame: Up to 4 weeks post-injection
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  Abdomen: Other | 1
  Chest/ thorax: Congenital disease/syndrome | 3
  Chest/ thorax: Infectious disease | 1
  Chest/ thorax: Malignant lesion | 1
  Chest/ thorax: No lesion/Normal | 6
  Chest/ thorax: Other | 2
  Brain: Other | 10
  Head/neck: Benign lesion | 1
  Head/neck: Malignant lesion | 1
  Head/neck: Other | 3
  Lymphatic system: Other | 1
  Pelvic area: Benign lesion | 1
  Pelvic area: Other | 1
  Retroperitoneal: Congenital disease/syndrome | 3
  Retroperitoneal: Malignant lesion | 1
  Retroperitoneal: Other | 3
  Spine: Malignant lesion | 1
  Spine: Other | 3
  Spine: Structural malformation | 1

31. Secondary Outcome: Number of Subjects With Change in Diagnosis From Unenhanced to Combined MRI
Description: The analysis value for change in diagnosis was recorded as "yes/no". Evaluation was done on pre- injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: FAS included all subjects who had combined unenhanced and enhanced image sets available regardless of any other protocol deviation.
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  No | 39
  Yes | 5

32. Secondary Outcome: Number of Subjects With Change in Diagnosis From Unenhanced to Combined MRI by Body Region
Description: The analysis value for change in diagnosis was recorded as "yes/no". Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 31
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  Abdomen: No | 1
  Abdomen: Yes | 0
  Brain: No | 20
  Brain: Yes | 1
  Chest/Thorax: No | 2
  Chest/Thorax: Yes | 0
  Head/Neck: No | 5
  Head/Neck: Yes | 0
  Lymphatic system: No | 1
  Lymphatic system: Yes | 0
  Pelvic area: No | 0
  Pelvic area: Yes | 2
  Retroperitoneal: No | 5
  Retroperitoneal: Yes | 2
  Spine: No | 5
  Spine: Yes | 0

33. Secondary Outcome: Number of Subjects With Change in Diagnosis From Unenhanced MRI to Final Diagnosis
Description: as for outcome 31
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 31
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  No | 33
  Yes | 11

34. Secondary Outcome: Number of Subjects With Change in Diagnosis From Unenhanced MRI to Final Diagnosis by Body Region
Description: as for outcome 32
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 31
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  Abdomen: No | 1
  Abdomen: Yes | 0
  Brain: No | 17
  Brain: Yes | 4
  Chest/Thorax: No | 1
  Chest/Thorax: Yes | 1
  Head/Neck: No | 4
  Head/Neck: Yes | 1
  Lymphatic system: No | 0
  Lymphatic system: Yes | 1
  Pelvic area: No | 1
  Pelvic area: Yes | 1
  Retroperitoneal: No | 5
  Retroperitoneal: Yes | 2
  Spine: No | 4
  Spine: Yes | 1

35. Secondary Outcome: Number of Subjects With Change in Diagnosis From Combined MRI to Final Diagnosis
Description: as for outcome 31
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 31
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  No | 32
  Yes | 12

36. Secondary Outcome: Number of Subjects With Change in Diagnosis From Combined MRI to Final Diagnosis by Body Region
Description: as for outcome 32
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 31
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  Abdomen: No | 1
  Abdomen: Yes | 0
  Brain: No | 16
  Brain: Yes | 5
  Chest/Thorax: No | 1
  Chest/Thorax: Yes | 1
  Head/Neck: No | 4
  Head/Neck: Yes | 1
  Lymphatic system: No | 0
  Lymphatic system: Yes | 1
  Pelvic area: No | 1
  Pelvic area: Yes | 1
  Retroperitoneal: No | 5
  Retroperitoneal: Yes | 2
  Spine: No | 4
  Spine: Yes | 1

37. Secondary Outcome: Number of Subjects With Change in Management From Unenhanced to Combined MRI
Description: The subject management was indicated based on the unenhanced images alone. The analysis value for change in subject management was recorded as "yes/no". Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 31
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  No | 36
  Yes | 8

38. Secondary Outcome: Number of Subjects With Change in Management From Unenhanced to Combined MRI by Body Region
Description: The subject management was indicated based on the unenhanced images alone. The analysis value for change in subject management was recorded as "yes/no". Results per body regions were reported. Evaluation was done on pre-injection and combined (pre- and post-injection) images.
Time Frame: Images were taken pre-injection and post-injection (within about 15 minutes)
Population: as for outcome 31
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  Abdomen: No | 1
  Abdomen: Yes | 0
  Brain: No | 19
  Brain: Yes | 2
  Chest/Thorax: No | 2
  Chest/Thorax: Yes | 0
  Head/Neck: No | 5
  Head/Neck: Yes | 0
  Lymphatic system: No | 1
  Lymphatic system: Yes | 0
  Pelvic area: No | 0
  Pelvic area: Yes | 2
  Retroperitoneal: No | 3
  Retroperitoneal: Yes | 4
  Spine: No | 5
  Spine: Yes | 0

39. Secondary Outcome: Number of Subjects With Clinically Significant Abnormal Laboratory Values
Description: Change in post-injection test values, such as resulting in a change in subject management or which were not the result of laboratory error and were considered clinically significant by the investigator was reported.
Time Frame: Baseline (not exceeding 24 hours before Gadobutrol injection) up to 24 hours post injection
Population: Safety Analysis Set (SAF) included all subjects who received any amount of gadobutrol.
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects | 0

40. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) Prior to Gadobutrol Injection
Description: eGFR was calculated based on the Schwartz formula with blood sampling for serum creatinine (Scr) not exceeding 14 days prior to gadobutrol injection. Otherwise, the eGFR was obtained from the original Schwartz formula: eGFR = k * height / Scr where k = 0.45 in term newborn infants < 1 year of age, and k = 0.55 in children up to 13 years of age. If Scr was measured by an enzymatic creatinine method that had been calibrated to be traceable to Isotope dilution mass spectroscopy (IDMS), the updated Schwartz formula was used: eGFR = 0.413*height/Scr.
Time Frame: Before gadobutrol injection
Population: SAF included all subjects who received any amount of gadobutrol. Here "n" included subjects who were evaluable at specified age group.
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 square
Arm/Group | Overall Study
Number analyzed (Participants) | 44
milliliter/minute/1.73 square
  < 1 month (n=5) | 61.8 (19.2)
  1 to < 2 months (n=4) | 91.7 (24.8)
  2 to < 6 months (n=9) | 136.3 (67.1)
  6 to < 12 months (n=11) | 115.2 (45.9)
  12 to < 24 months (n=15) | 150.4 (33.9)

41. Other Pre Specified Outcome: Number of Subjects With Drug Related Serious and Non- Serious Adverse Events
Description: An Adverse Event (AE) was any untoward medical occurrence in a subject who received study drug. A Serious AE (SAE) was an AE resulting in death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly, or deemed significant for any other reason. The drug-relatedness of AEs was determined by the Investigator based on his/her clinical decision based on all available information, and was based on the question whether there was a "reasonable causal relationship" to the study treatment.
Time Frame: From baseline to approximately 7 days after injection
Population: SAF included all subjects who received any amount of gadobutrol.
Measure: Number; unit: subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 44
subjects
  Any study drug-related AE | 1
  Any study drug-related SAE | 0

ADVERSE EVENTS:
Time Frame: From baseline to approximately 7 days after injection.
Description: (S)AEs detailed below are both drug-unrelated and related. One non-serious adverse drug reaction (ADR) of Vomiting was reported in one subject (2.3%). Please refer to "other pre-specified endpoint 41" under "outcome measures.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 3/44
Other Adverse Events (participants affected / at risk) | 17/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=44)
Infected cyst (Infections and infestations) | 1 (1)
Subdural empyema (Infections and infestations) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=44)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Catheter site erythema (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Nasopharyngitis (Infections and infestations) | 3 (4)
Rash pustular (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2)
Body temperature increased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Convulsion (Nervous system disorders) | 1 (2)
Urine odour abnormal (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Results for Typical PK parameters were provided by the median value of the population together with the min-max range (individual PK). Typical PK parameter as described in study protocol was reflected by the Median PK parameter in the study report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is interested in the publication of the results of every study it performs. All relevant aspects regarding publication will be part of the contract between the sponsor and the investigator/institution.